CLINICAL TRIAL: NCT04451538
Title: Impact of Perioperative Nutritional Intervention on Perioperative Outcomes of Elderly Patients Having Hip Fracture Surgery: A Randomized Control Trial
Brief Title: Nutritional Intervention and Outcomes in Elderly After Hip Fracture Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was stopped prematurely due to slow recruitment.
Sponsor: Peking University First Hospital (Other)
Collaborators: The Forth Medical Center of PLA General Hospital (Unknown); Tianjin Orthopedic Hospital (Unknown)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-322
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Elderly Patients; Malnutrition; Hip Fractures; Nutritional Intervention; Perioperative Outcomes; Survival
Keywords: Elderly patients; Malnutrition; Hip Fractures; Nutritional intervention; Perioperative outcomes; Long-term survival
MeSH Terms: conditions — Malnutrition; Hip Fractures | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nutritional intervention group (Experimental): Supplemental nutritional support is provided in addition to normal diet during the perioperative period (five days from pre- to postoperative phase). For non-diabetic patients, ENSURE is provided (Abbott; 112.6 g [12 spoon, 500 kcal]/day, twice a day); for diabetic patients, GLUCERNA SR is provided (Abbott; 104 g [12 spoon, 440 kcal]/day, twice a day).
  Interventions: Dietary Supplement: Nutritional intervention group
- Control group (Placebo Comparator): Supplemental nutritional support is not provided in addition to normal diet during the perioperative period (five days from pre- to postoperative phase).
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Nutritional intervention group — Supplemental nutritional support is provided in addition to normal diet during the perioperative period (five days from pre- to postoperative phase). For non-diabetic patients, ENSURE is provided (Abbott; 112.6 g (12 spoons, 500 kcal)/day, twice a day); for diabetic patients, GLUCERNA SR is provided (Abbott; 104 g [12 spoons, 440 kcal]/day, twice a day).
  Arms: Nutritional intervention group
Dietary Supplement: Control group — Supplemental nutritional support is not provided in addition to normal diet during the perioperative period (five days from pre- to postoperative phase).
  Arms: Control group

SUMMARY:
Hip fracture is one of the most frequently occurred injury in the elderly and usually requires surgical treatment. Malnutrition is common in elderly patients with hip fracture and is associated with worse outcomes. This study is designed to test the hypothesize that, in elderly patients with malnutrition or at risk of malnutrition and scheduled for hip-fracture surgery, perioperative nutritional intervention may reduce early complications and improve long-term survival.

DETAILED DESCRIPTION:
Elderly patients with hip fracture have a high rate of malnutrition. In a cohort study of hip fracture patients aged 70 years or older, 18.8% have malnutrition and 44.6% are at risk of malnutrition. Increasing evidence suggest that preoperative nutritional status has a significant impact on clinical outcomes of elderly patients following surgery. For example, preoperative malnutrition or risk of malnutrition is associated with increased delirium, increased non-delirium complications, prolonged hospital stay, high mortality, and even worse long-term survival after surgery. We speculate that perioperative nutritional intervention may reduce postoperative delirium and improve early and long-term clinical outcomes in elderly hip-fracture patients. The purpose of this study is to observe the effect of perioperative nutritional intervention on early postoperative delirium and complications as well as long-term survival in the patients with malnutrition or at risk of malnutrition who are scheduled for hip-fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years old;
* Hospitalized for hip fracture, scheduled to undergo hip-fracture surgery within 48 hours;
* Classified as malnutrition or at risk of malnutrition according to the short form mini-nutrition assessment (MNA-SF);
* Provide written informed consents.

Exclusion Criteria:

* Pathological fracture;
* History of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis before surgery;
* Unable to communicate due to coma, severe dementia, or language barrier;
* Unable to eat due to any disease in the gastrointestinal system;
* Severe hepatic dysfunction (Child-Pugh class C), renal failure (requirement of renal replacement therapy), respiratory failure (requirement of respiratory support), cardiac insufficiency (New York Heart Association classification ≥IV), or American Socisty of Anesthesiologists classification ≥IV;
* Preexisting organ injury before surgery (delirium, acute kidney injury, myocardial injury, etc.);
* Other conditions that are considered unsuitable for study participation.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium or non-delirium complications after surgery | Up to 30 days after surgery
  Delirium is assessed twice daily with Confusion Assessment Method (CAM) or CAM for the Intensive Care Unit (CAM-ICU) during the first 5 days after surgery. Non-delirium complications indicate newly occurred conditions (other than delirium) that are harmful to patients' recovery and required therapeutic intervention within 30 days after surgery.

SECONDARY OUTCOMES:
Intensive care unit admission after surgery | Within 24 hours after surgery
  Intensive care unit admission after surgery
Length of intensive care unit stay after surgery | Up to 30 days after surgery
  Length of intensive care unit stay after surgery
Incidence of organ injury within 5 days after surgery | Up to 5 days after surgery
  Organ injury includes delirium (assessed with CAM/CAM-ICU), acute kidney injury (assessed according to KDIGO [Kidney Disease: Improving Global Outcomes] Criteria), and myocardial injury (cardiac troponin I higher than upper normal limit).
Incidence of non-delirium complications after surgery | Up to 30 days after surgery
  Non-delirium complications indicate newly occurred conditions (other than delirium) that are harmful to patients' recovery and required therapeutic intervention within 30 days after surgery.
Length of hospital stay after surgery | Up to 30 days after surgery.
  Length of hospital stay after surgery
Cognitive function at 30 days after surgery | At 30 days after surgery.
  Cognitive function is assessed with the Modified Telephone Interview for Cognitive Status (TICS-m) which is a 12-item questionnaire that verbally assesses global cognitive function via telephone. The score ranges from 0 to 50, with higher score indicating better function.
Quality of life at 30 days after surgery | At 30 days after surgery.
  Quality of life is assessed with the World Health Organization Quality of Life brief version (WHOQOL-BREF) which is a 24-item questionnaire that assesses the quality of life in physical, psychological, social relationship and environmental domains. The score ranges from 0 to 100 for each domain, with higher score indicating better function.

OTHER OUTCOMES:
Pain intensity. | During the first 5 days after surgery
  Pain intensity is assessed twice daily (8:00-10:00, 18:00-20:00) with the numeric rating scale (NRS; which is an 11-point scale whereas 0=no pain and 10=the worst pain).
Subjective sleep quality. | During the first 5 days after surgery
  Subjective sleep quality is assessed once daily (8:00-10:00) with the numeric rating scale (NRS; which is an 11-point scale whereas 0=the best sleep and 10=the worst sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fourth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Tianjin Orthopedic Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brauer CA, Coca-Perraillon M, Cutler DM, Rosen AB. Incidence and mortality of hip fractures in the United States. JAMA. 2009 Oct 14;302(14):1573-9. doi: 10.1001/jama.2009.1462. PMID 19826027
- [Background] Membership of the Working Party; Griffiths R, Alper J, Beckingsale A, Goldhill D, Heyburn G, Holloway J, Leaper E, Parker M, Ridgway S, White S, Wiese M, Wilson I. Management of proximal femoral fractures 2011: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2012 Jan;67(1):85-98. doi: 10.1111/j.1365-2044.2011.06957.x. PMID 22150501
- [Background] Mak JC, Cameron ID, March LM; National Health and Medical Research Council. Evidence-based guidelines for the management of hip fractures in older persons: an update. Med J Aust. 2010 Jan 4;192(1):37-41. doi: 10.5694/j.1326-5377.2010.tb03400.x. PMID 20047547
- [Background] Cram P, Lu X, Kaboli PJ, Vaughan-Sarrazin MS, Cai X, Wolf BR, Li Y. Clinical characteristics and outcomes of Medicare patients undergoing total hip arthroplasty, 1991-2008. JAMA. 2011 Apr 20;305(15):1560-7. doi: 10.1001/jama.2011.478. PMID 21505134
- [Background] Bottle A, Aylin P. Mortality associated with delay in operation after hip fracture: observational study. BMJ. 2006 Apr 22;332(7547):947-51. doi: 10.1136/bmj.38790.468519.55. Epub 2006 Mar 22. PMID 16554334
- [Background] Shiga T, Wajima Z, Ohe Y. Is operative delay associated with increased mortality of hip fracture patients? Systematic review, meta-analysis, and meta-regression. Can J Anaesth. 2008 Mar;55(3):146-54. doi: 10.1007/BF03016088. PMID 18310624
- [Background] Moja L, Piatti A, Pecoraro V, Ricci C, Virgili G, Salanti G, Germagnoli L, Liberati A, Banfi G. Timing matters in hip fracture surgery: patients operated within 48 hours have better outcomes. A meta-analysis and meta-regression of over 190,000 patients. PLoS One. 2012;7(10):e46175. doi: 10.1371/journal.pone.0046175. Epub 2012 Oct 3. PMID 23056256
- [Background] Espinosa KA, Gelvez AG, Torres LP, Garcia MF, Pena OR. Pre-operative factors associated with increased mortality in elderly patients with a hip fracture: A cohort study in a developing country. Injury. 2018 Jun;49(6):1162-1168. doi: 10.1016/j.injury.2018.04.007. Epub 2018 Apr 13. PMID 29674111
- [Background] Smith T, Pelpola K, Ball M, Ong A, Myint PK. Pre-operative indicators for mortality following hip fracture surgery: a systematic review and meta-analysis. Age Ageing. 2014 Jul;43(4):464-71. doi: 10.1093/ageing/afu065. Epub 2014 Jun 3. PMID 24895018
- [Background] Malafarina V, Reginster JY, Cabrerizo S, Bruyere O, Kanis JA, Martinez JA, Zulet MA. Nutritional Status and Nutritional Treatment Are Related to Outcomes and Mortality in Older Adults with Hip Fracture. Nutrients. 2018 Apr 30;10(5):555. doi: 10.3390/nu10050555. PMID 29710860
- [Background] Yang Y, Zhao X, Dong T, Yang Z, Zhang Q, Zhang Y. Risk factors for postoperative delirium following hip fracture repair in elderly patients: a systematic review and meta-analysis. Aging Clin Exp Res. 2017 Apr;29(2):115-126. doi: 10.1007/s40520-016-0541-6. Epub 2016 Feb 12. PMID 26873816
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702
- [Background] McDaniel M, Brudney C. Postoperative delirium: etiology and management. Curr Opin Crit Care. 2012 Aug;18(4):372-6. doi: 10.1097/MCC.0b013e3283557211. PMID 22732435
- [Background] Lat I, McMillian W, Taylor S, Janzen JM, Papadopoulos S, Korth L, Ehtisham A, Nold J, Agarwal S, Azocar R, Burke P. The impact of delirium on clinical outcomes in mechanically ventilated surgical and trauma patients. Crit Care Med. 2009 Jun;37(6):1898-905. doi: 10.1097/CCM.0b013e31819ffe38. PMID 19384221
- [Background] Quinlan N, Rudolph JL. Postoperative delirium and functional decline after noncardiac surgery. J Am Geriatr Soc. 2011 Nov;59 Suppl 2:S301-4. doi: 10.1111/j.1532-5415.2011.03679.x. PMID 22091577
- [Background] Lescot T, Karvellas CJ, Chaudhury P, Tchervenkov J, Paraskevas S, Barkun J, Metrakos P, Goldberg P, Magder S. Postoperative delirium in the intensive care unit predicts worse outcomes in liver transplant recipients. Can J Gastroenterol. 2013 Apr;27(4):207-12. doi: 10.1155/2013/289185. PMID 23616958
- [Background] Abelha FJ, Luis C, Veiga D, Parente D, Fernandes V, Santos P, Botelho M, Santos A, Santos C. Outcome and quality of life in patients with postoperative delirium during an ICU stay following major surgery. Crit Care. 2013 Oct 29;17(5):R257. doi: 10.1186/cc13084. PMID 24168808
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Stuck A, Clark MJ, Connelly CD. Preventing intensive care unit delirium: a patient-centered approach to reducing sleep disruption. Dimens Crit Care Nurs. 2011 Nov-Dec;30(6):315-20. doi: 10.1097/DCC.0b013e31822fa97c. PMID 21983504
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259
- [Background] Smith TO, Cooper A, Peryer G, Griffiths R, Fox C, Cross J. Factors predicting incidence of post-operative delirium in older people following hip fracture surgery: a systematic review and meta-analysis. Int J Geriatr Psychiatry. 2017 Apr;32(4):386-396. doi: 10.1002/gps.4655. Epub 2017 Jan 17. PMID 28093812
- [Background] Oh ES, Li M, Fafowora TM, Inouye SK, Chen CH, Rosman LM, Lyketsos CG, Sieber FE, Puhan MA. Preoperative risk factors for postoperative delirium following hip fracture repair: a systematic review. Int J Geriatr Psychiatry. 2015 Sep;30(9):900-10. doi: 10.1002/gps.4233. Epub 2014 Dec 11. PMID 25503071
- [Background] Nuotio M, Tuominen P, Luukkaala T. Association of nutritional status as measured by the Mini-Nutritional Assessment Short Form with changes in mobility, institutionalization and death after hip fracture. Eur J Clin Nutr. 2016 Mar;70(3):393-8. doi: 10.1038/ejcn.2015.174. Epub 2015 Oct 21. PMID 26486304
- [Background] Guyonnet S, Rolland Y. Screening for Malnutrition in Older People. Clin Geriatr Med. 2015 Aug;31(3):429-37. doi: 10.1016/j.cger.2015.04.009. Epub 2015 May 13. PMID 26195101
- [Background] Deutz NE, Matheson EM, Matarese LE, Luo M, Baggs GE, Nelson JL, Hegazi RA, Tappenden KA, Ziegler TR; NOURISH Study Group. Readmission and mortality in malnourished, older, hospitalized adults treated with a specialized oral nutritional supplement: A randomized clinical trial. Clin Nutr. 2016 Feb;35(1):18-26. doi: 10.1016/j.clnu.2015.12.010. Epub 2016 Jan 18. PMID 26797412
- [Background] Zhang Y, Shan GJ, Zhang YX, Cao SJ, Zhu SN, Li HJ, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) Investigators. Preoperative vitamin D deficiency increases the risk of postoperative cognitive dysfunction: a predefined exploratory sub-analysis. Acta Anaesthesiol Scand. 2018 Aug;62(7):924-935. doi: 10.1111/aas.13116. Epub 2018 Mar 26. PMID 29578249
- [Background] Zhang DF, Su X, Meng ZT, Cui F, Li HL, Wang DX, Li XY. Preoperative severe hypoalbuminemia is associated with an increased risk of postoperative delirium in elderly patients: Results of a secondary analysis. J Crit Care. 2018 Apr;44:45-50. doi: 10.1016/j.jcrc.2017.09.182. Epub 2017 Sep 29. PMID 29055835
- [Background] Mazzola P, Ward L, Zazzetta S, Broggini V, Anzuini A, Valcarcel B, Brathwaite JS, Pasinetti GM, Bellelli G, Annoni G. Association Between Preoperative Malnutrition and Postoperative Delirium After Hip Fracture Surgery in Older Adults. J Am Geriatr Soc. 2017 Jun;65(6):1222-1228. doi: 10.1111/jgs.14764. Epub 2017 Mar 6. PMID 28263371
- [Background] Olofsson B, Stenvall M, Lundstrom M, Svensson O, Gustafson Y. Malnutrition in hip fracture patients: an intervention study. J Clin Nurs. 2007 Nov;16(11):2027-38. doi: 10.1111/j.1365-2702.2006.01864.x. Epub 2007 Apr 5. PMID 17419798
- [Background] Avenell A, Smith TO, Curtain JP, Mak JC, Myint PK. Nutritional supplementation for hip fracture aftercare in older people. Cochrane Database Syst Rev. 2016 Nov 30;11(11):CD001880. doi: 10.1002/14651858.CD001880.pub6. PMID 27898998
- [Background] Griffiths R, Beech F, Brown A, Dhesi J, Foo I, Goodall J, Harrop-Griffiths W, Jameson J, Love N, Pappenheim K, White S; Association of Anesthetists of Great Britain and Ireland. Peri-operative care of the elderly 2014: Association of Anaesthetists of Great Britain and Ireland. Anaesthesia. 2014 Jan;69 Suppl 1:81-98. doi: 10.1111/anae.12524. PMID 24303864
- [Background] Rubenstein LZ, Harker JO, Salva A, Guigoz Y, Vellas B. Screening for undernutrition in geriatric practice: developing the short-form mini-nutritional assessment (MNA-SF). J Gerontol A Biol Sci Med Sci. 2001 Jun;56(6):M366-72. doi: 10.1093/gerona/56.6.m366. PMID 11382797
- [Background] Inoue T, Misu S, Tanaka T, Kakehi T, Ono R. Acute phase nutritional screening tool associated with functional outcomes of hip fracture patients: A longitudinal study to compare MNA-SF, MUST, NRS-2002 and GNRI. Clin Nutr. 2019 Feb;38(1):220-226. doi: 10.1016/j.clnu.2018.01.030. Epub 2018 Feb 15. PMID 29456030
- [Background] O'Hara DA, Duff A, Berlin JA, Poses RM, Lawrence VA, Huber EC, Noveck H, Strom BL, Carson JL. The effect of anesthetic technique on postoperative outcomes in hip fracture repair. Anesthesiology. 2000 Apr;92(4):947-57. doi: 10.1097/00000542-200004000-00011. PMID 10754613
- [Background] Neuman MD, Silber JH, Elkassabany NM, Ludwig JM, Fleisher LA. Comparative effectiveness of regional versus general anesthesia for hip fracture surgery in adults. Anesthesiology. 2012 Jul;117(1):72-92. doi: 10.1097/ALN.0b013e3182545e7c. PMID 22713634
- [Background] Fields AC, Dieterich JD, Buterbaugh K, Moucha CS. Short-term complications in hip fracture surgery using spinal versus general anaesthesia. Injury. 2015 Apr;46(4):719-23. doi: 10.1016/j.injury.2015.02.002. Epub 2015 Feb 11. PMID 25704139
- [Background] Neuman MD, Rosenbaum PR, Ludwig JM, Zubizarreta JR, Silber JH. Anesthesia technique, mortality, and length of stay after hip fracture surgery. JAMA. 2014 Jun 25;311(24):2508-17. doi: 10.1001/jama.2014.6499. PMID 25058085
- [Background] Patorno E, Neuman MD, Schneeweiss S, Mogun H, Bateman BT. Comparative safety of anesthetic type for hip fracture surgery in adults: retrospective cohort study. BMJ. 2014 Jun 27;348:g4022. doi: 10.1136/bmj.g4022. PMID 24972901
- [Background] Robinson TN, Walston JD, Brummel NE, Deiner S, Brown CH 4th, Kennedy M, Hurria A. Frailty for Surgeons: Review of a National Institute on Aging Conference on Frailty for Specialists. J Am Coll Surg. 2015 Dec;221(6):1083-92. doi: 10.1016/j.jamcollsurg.2015.08.428. Epub 2015 Sep 11. No abstract available. PMID 26422746